CLINICAL TRIAL: NCT00004089
Title: A Multicenter Phase II Study of Intensified Concomitant Chemoradiotherapy for Patients With Anaplastic Thyroid Cancer
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Previously Untreated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU V96N3; NU-V96N3; UCCRC-08200; NCI-G99-1580
Record Dates: First submitted 1999-12-10; First posted 2004-09-14 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2011-01

CONDITIONS: Head and Neck Cancer
Keywords: anaplastic thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Carcinoma, Anaplastic | interventions — Filgrastim; Fluorouracil; Hydroxyurea; Paclitaxel; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: fluorouracil
Drug: hydroxyurea
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have previously untreated anaplastic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the activity of chemotherapy with hyperfractionated radiotherapy in terms of complete and overall response rate, time to progression, pattern of failure, incidence of second primary tumors, and overall survival in patients with previously untreated anaplastic thyroid cancer.

OUTLINE: This is a multicenter study. Patients receive oral hydroxyurea every 12 hours on days 0-5, fluorouracil IV and paclitaxel IV continuously over days 1-5, and hyperfractionated radiotherapy twice daily on days 1-5. Patients receive filgrastim (G-CSF) subcutaneously daily on days 6-12. Treatment repeats every 2 weeks for 5 courses. Following completion of concurrent chemoradiotherapy, patients with no prior initial modified neck dissection who have residual macroscopic nodal disease or initially staged nodal disease with no evidence of residual disease undergo neck dissection. Patients with macroscopic residual disease at the primary site undergo complete excision of disease. Patients with any progressive disease or recurrence of disease undergo conventional surgical management. Patients are followed at 4-6 weeks, every 3 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 16-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed anaplastic thyroid cancer Metastatic disease allowed

PATIENT CHARACTERISTICS: Age: 15 to 80 Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Alkaline phosphatase no greater than 2 times normal Transaminases no greater than 2 times normal Renal: Not specified

PRIOR CONCURRENT THERAPY: Prior simple excision (e.g., transoral laser excision) of the primary lesion allowed if organ function preserved Prior modified neck dissection allowed

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merrill S. Kies, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois